CLINICAL TRIAL: NCT01548664
Title: The Utilization of Nintendo Wii™ in Outpatient Rehabilitation Following Total Knee Replacement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Manuel Gomez, MD, MSc. (Other)
Responsible Party: Sponsor-Investigator, Manuel Gomez, MD, MSc., Director of the Clinical Research Department, St. John's Rehab Hospital
Organization: St. John's Rehab Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-02
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Arthropathy of Knee Joint
Keywords: Total knee replacement; Outpatient; Randomized controlled trial; Video games

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nintendo Wii FitTM (Experimental): Fifteen minutes of gaming activity on the Wii Fit™ following each regularly scheduled 60 minute physiotherapy session, in a separate treatment area.
  Interventions: Other: Wii Fit
- Lower extremity exercise (Active Comparator): Fifteen minutes of lower extremity exercises that addressed balance, posture, weight shifting and strengthening were provided bilaterally, following each regularly scheduled 60 minute physiotherapy session, in a separate treatment area
  Interventions: Other: Lower Extremity Exercise

INTERVENTIONS:
Other: Wii Fit — 15 minutes of gaming activity on the Wii Fit™ following each regularly scheduled 60 minute physiotherapy session, in a separate treatment area.
  Other Names: Nintendo Wii Fit
  Arms: Nintendo Wii FitTM
Other: Lower Extremity Exercise — Fifteen minutes of lower extremity exercise that addressed balance, posture, weight shifting and strengthening provided bilaterally following each regularly scheduled 60 minute physiotherapy session, in a separate treatment area.
  Arms: Lower extremity exercise

SUMMARY:
The purpose of this study is to identify whether the utilization of the Nintendo Wii™ gaming system, as an adjunct to conventional outpatient rehabilitation therapy, influence outcomes of patients following total knee replacement (TKR). The investigators hypothesize that the Nintendo Wii™ gaming system has a positive influence in the outcomes of patients following TKR.

DETAILED DESCRIPTION:
The use of video games in rehabilitation is growing in popularity and frequency. The Nintendo Wii™ gaming system in particular, is gaining increased attention in the rehabilitation setting. There is currently very little evidence to support its clinical use. Canadian total knee replacement (TKR) rates have risen significantly in the past decade and its patient demographic has shifted to reflect a younger overall population. These changes indicate increased emphasis on TKR patients returning to higher levels of function and the potential need for new intervention options when caring for these patients. The Nintendo Wii™ Sports application has the potential to encourage standing, while participating in an interesting and engaging activity. The objective of this study is to determine whether the utilization of the Nintendo Wii™ gaming system, as an adjunct to standard outpatient rehabilitation therapy, influence outcomes of patients following total knee replacement.

Patients who consent to participate in this study will be randomized to either a control group which will receive 15 minutes of lower extremity exercise or a study group which will receive 15 minutes of gaming activity on the Wii Fit™. Both control and study interventions will be provided following each regularly scheduled 60 minute physiotherapy session, in a separate treatment area. The Nintendo Wii™ console and its accompanying Wii™ Sports game will be utilized for the purposes of this study. To minimize rotational movement and therefore the risk of injury following total knee replacement, only the tennis and bowling games will be used. It will be required that these games are played in standing position. Without including the time required for start-up, each session of Nintendo Wii™ game activity will be 15 minutes in duration, and will be provided twice weekly.

Recovery status will be measured in all participants on admission, and every 2 weeks until discharge, an expected average of 5 weeks. A combination of self-administered questionnaires, objective and subjective outcome measures will be used to measure function (2 Minute Walk Test, Lower Extremity Functional Scale) range of motion (Goniometry), pain (Numeric Pain Rating Scale) and satisfaction with therapy services. Change within each measure will be statistically analyzed to detect whether a significant difference exists between control and study groups. It is projected that 60 patients will be recruited for this study. Patients in the study group could potentially benefit from increased improvements in pain, physical status, function, and satisfaction at the completion of their outpatient rehabilitation therapy program.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with full lower extremity weight bearing
* Requiring physiotherapy treatment twice weekly for Total Knee Arthroplasty rehabilitation.

Exclusion Criteria:

* Individuals with visual impairments
* Active painful osteoarthritis in the contralateral lower extremity
* Patients with uncorrected visual impairments
* English language barriers or impairments to their ability to follow instruction.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Length of outpatient rehab stay (LOS) | From admission to discharge, an expected average of 5 weeks.
  Days from admission to discharge from the outpatient rehabilitation program

SECONDARY OUTCOMES:
Lower Extremity Functional Scale | From admission to discharge, an expected average of 5 weeks.
  The Lower Extremity Functional Scale will be administer on the first study visit and every two weeks until discharged from outpatient physiotherapy services by their treating clinician.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Fung, BSc, MSc.PT., Principal Investigator — St. John's Rehab Hospital
Locations (1):
- St. John's Rehab Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Fung V, Ho A, Shaffer J, Gomez M. The Utilization of Nintendo Wii Fit in the Rehabilitation of Outpatients Following Total Knee Replacements: Preliminary Results of a Randomized Controlled Trial. Archives of Physical Medicine and Rehabilitation 91(10): e37, 2010.
- [Derived] Fung V, Ho A, Shaffer J, Chung E, Gomez M. Use of Nintendo Wii Fit in the rehabilitation of outpatients following total knee replacement: a preliminary randomised controlled trial. Physiotherapy. 2012 Sep;98(3):183-8. doi: 10.1016/j.physio.2012.04.001. Epub 2012 Jul 10. PMID 22898573